CLINICAL TRIAL: NCT03172702
Title: A Phase 3 Multicenter Open-label Maintenance Study to Investigate the Long-term Safety of ZS (Sodium Zirconium Cyclosilicate) in Japanese Subjects With Hyperkalemia
Brief Title: Open-label Safety of Sodium Zirconium Cyclosilicate for up to 12 Months in Japanese Subjects With Hyperkalemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: D9482C00001
Record Dates: First submitted 2017-05-22; First posted 2017-06-01 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sodium Zirconium Cyclosilicate (Experimental): Correction Phase Dosing: Sodium Zirconium Cyclosilicate 10 g three times daily (TID) from 24 to 72 Extended Dosing: Sodium Zirconium Cyclosilicate 5 g once daily (QD). Sodium Zirconium Cyclosilicate dose increased or decreased in increments/decrements of 5 g QD up to a maximum of 15 g QD or a minimum of 5 g every other day (QOD) (or 2.5 g QD) based on i-STAT potassium measurements up to 12 months.
  Interventions: Drug: Zirconium Cyclosilicate

INTERVENTIONS:
Drug: Zirconium Cyclosilicate — Correction Phase Dosing: Sodium Zirconium Cyclosilicate 10 g three times daily (TID) from 24 to 72 Extended Dosing: Sodium Zirconium Cyclosilicate 5 g once daily (QD). Sodium Zirconium Cyclosilicate dose increased or decreased in increments/decrements of 5 g QD up to a maximum of 15 g QD or a minimum of 5 g every other day (QOD) (or 2.5 g QD) based on i-STAT potassium measurements up to 12 months.
  Other Names: ZS

SUMMARY:
The Open-Label Maintenance Study contains an Correction Phase, in which subjects will be dosed with ZS 10 g three times daily (tid) for 24 to 72 hours, followed by a 12-month long-term Maintenance Phase.

DETAILED DESCRIPTION:
The study will start with the screening period, and all baseline parameters should be measured/collected up to 1 day prior to administration of first dose of study drug on Correction Phase Day 1. Subjects with 2 consecutive i-STAT potassium values ≥ 5.1 mmol/L will enter the Correction Phase and receive ZS 10 g TID for up to 72 hours, depending on potassium values. Once normokalemia (i-STAT potassium between 3.5 and 5.0 mmol/L, inclusive) is restored (whether after 24, 48 or 72 hours), subjects will be entered into the Maintenance Phase to be dosed with ZS at a starting dose of 5 g QD. Potassium (i-STAT and Central Laboratory) will be measured Days 1, 2, 5, 12, 19 and 26 throughout the first month of study and every 4 weeks thereafter until Day 362 (Visit 23) then patients will be required to complete the EOS visit which is 7±1 days after the last administration of study medication. For patients who do not enter the Maintenance Phase the last visit will be 7±1 day after the last treatment dose in the Correction Phase. The total expected study duration for an individual patient is approximately 53-54 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Patients aged ≥18. For patients aged <20 years, a written informed consent should be obtained from the patient and his or her legally acceptable representative.
* Two consecutive i-STAT potassium values, measured 60-minutes (± 15 minutes) apart, both ≥ 5.1 mmol/L and measured within 1 day before the first dose of ZS on Correction Phase Study Day 1.
* Patients who are on peritoneal dialysis (PD) can be enrolled if their SK level is ≥5.5 and ≤ 6.5 mmol/L in two consecutive i-STAT potassium evaluation at least 24 hours apart before Day 1 (in each evaluation, two i-STAT potassium measurements at least 1 hour apart are required). i-STAT potassium measurement should be performed in the morning before breakfast and in the evening before dinner in PD patients on continuous ambulatory peritoneal dialysis (CAPD) and automated peritoneal dialysis (APD), respectively.
* Women of childbearing potential must be using 2 forms of medically acceptable contraception (at least 1 barrier method) and have a negative pregnancy test within 1 day prior to the first dose of ZS on Correction Phase Study Day 1. Women who are surgically sterile or those who are postmenopausal for at least 1 year are not considered to be of childbearing potential.

Exclusion Criteria:

* Patients treated with lactulose, rifaxan (rifaximin), or other non-absorbed antibiotics for hyperammonemia within 7 days prior to first dose of ZS.
* Patients treated with resins (such as sevelamer hydrochloride, sodium polystyrene sulfonate [SPS; e.g. Kayexalate®] or calcium polystyrene sulfonate [CPS]), calcium acetate, calcium carbonate, or lanthanum carbonate, within 7 days prior to the first dose of study drug. Washout of SPS and CPS for 7 days (or longer) prior to the first dose of ZS is allowed, if termination of CPS or SPS is judged to be clinically acceptable by the investigator. Documented informed consent has to be obtained prior to the washout.
* Patients with a life expectancy of less than 12 months
* Female patients who are pregnant, lactating, or planning to become pregnant
* Patients who have an active or history of diabetic ketoacidosis
* Known hypersensitivity or previous anaphylaxis to ZS or to components thereof
* Treatment with a drug or device within the last 30 days that has not received regulatory approval at the time of study entry.
* Patients with cardiac arrhythmias that require immediate treatment
* Hemodialysis patients (including those who are on both PD and hemodialysis [HD])
* Patients who have been on PD less than 6 months or more than 6 months with a history of hypokalemia within 6 months before Correction Phase Day 1
* Documented Glomerular Filtration Rate (GFR) < 15 mL/min within 90 days prior to study entry (Non peritoneal dialysis (PD) patients only)
* If patients joined ZS study in the past, the patients cannot join this study within the last 30 days of the last study drug administration day.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- Japan (37):
  - Research Site, Akashi-shi
  - Research Site, Amagasaki-shi
  - Research Site, Chiba
  - Research Site, Chiyoda-ku
  - Research Site, Chūōku
  - Research Site, Funabashi-shi
  - Research Site, Hanyu-shi
  - Research Site, Higashiibaraki-gun
  - Research Site, Hitachi-Naka
  - Research Site, Ina-shi
  - Research Site, Kagoshima
  - Research Site, Kahoku-gun
  - Research Site, Kamakura-shi
  - Research Site, Kasuga-shi
  - Research Site, Kasugai-shi
  - Research Site, Kawachinagano-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Kochi
  - Research Site, Koga-shi
  - Research Site, Kumamoto
  - Research Site, Matsudo-shi
  - Research Site, Matsuyama
  - Research Site, Minokamo-shi
  - Research Site, Mito
  - Research Site, Nagoya
  - Research Site, Naka
  - Research Site, Omura-shi
  - Research Site, Onomichi-shi
  - Research Site, Osaka
  - Research Site, Shimajiri-gun
  - Research Site, Shizuoka
  - Research Site, Toride-shi
  - Research Site, Toshima-ku
  - Research Site, Toyohashi
  - Research Site, Yakushi
  - Research Site, Yotsukaido-shi

REFERENCES:
- [Derived] Kashihara N, Yamasaki Y, Osonoi T, Harada H, Shibagaki Y, Zhao J, Kim H, Yajima T, Sarai N. A phase 3 multicenter open-label maintenance study to investigate the long-term safety of sodium zirconium cyclosilicate in Japanese subjects with hyperkalemia. Clin Exp Nephrol. 2021 Feb;25(2):140-149. doi: 10.1007/s10157-020-01972-y. Epub 2020 Oct 24. PMID 33098526
- See also: D9482C0000 redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9482C00001&attachmentIdentifier=98c4b9be-0b01-4391-a1da-8544ff12da15&fileName=D9482C00001_CSP_redacted.pdf&versionIdentifier=
- See also: D9482C00001 redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9482C00001&attachmentIdentifier=6fcba409-a47f-4c13-a467-f36a2e9f9e10&fileName=D9482C00001_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese patients with hyperkalemia were recruited to this open-label, single-arm study with a flexible dosing regimen conducted in 44 study centers in Japan. First patient enrolled in September 2017; last patient completed in July 2019.
Pre-assignment Details: For inclusion, patients were required to have 2 consecutive iSTAT (portable blood analyzer) potassium values, measured 60 minutes apart, both ≥5.1 millimole per liter (mmol/L) and measured within 1 day before the first dose of sodium zirconium cyclosilicate (ZS) on Correction Phase (CP) Day 1.
Groups:
- Sodium Zirconium Cyclosilicate: CP (up to 3 days):
  Patients received 10 grams (g) ZS three times daily (TID) for a maximum of 72 hours. If a patient became normokalemic (iSTAT potassium ≥3.5 and ≤5.0 mmol/L) after 24, 48 or 72 hours they progressed to the Maintenance Phase (MP).
  MP (up to 12 months):
  Patients received a starting dose of 5 g ZS once daily (QD) and based on the iSTAT potassium measurements the ZS dose could be increased to 10 g or 15 g QD or decreased to 5 g once every other day (QOD) or 2.5 g QD.
Period: Overall Study
Arm/Group | Sodium Zirconium Cyclosilicate
Started (Started the CP) | 150
Received Treatment in CP | 150
Received Treatment in MP | 150
Completed (Completed treatment in the MP) | 122
Not Completed | 28
Not completed — Adverse Event | 9
Not completed — Death | 2
Not completed — Study-specific Withdrawal Criteria | 10
Not completed — Withdrawal by Subject | 5
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- Sodium Zirconium Cyclosilicate: CP (up to 3 days):
  Patients received 10 g ZS TID for a maximum of 72 hours.
  MP (up to 12 months):
  Patients received a starting dose of 5 g ZS QD which could be increased to 10 g or 15 g QD or decreased to 5 g QOD or 2.5 g QD.
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced Adverse Events (AEs) in the MP
Description: The number of patients who experienced any AE, including those which were serious (SAE), had an outcome of death, were severe, led to discontinuation of ZS or were causally related to ZS are presented for the MP. AEs of special interest are also presented, including oedema-related AEs, cardiac failure and hypertension.
Time Frame: First MP dose up to 1 day (2 days for QOD regimen) after last MP dose.
Population: The safety analysis set for the MP (SAF-MP) included all patients treated with at least 1 dose of MP ZS and who had any MP safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Participants
  Any AE | 131
  Any AE with outcome death | 2
  Any SAE | 27
  Any severe AE | 9
  Any AE leading to ZS discontinuation | 12
  Any causally related AE | 30
  Oedema-related AE | 31
  Cardiac failure | 10
  Hypertension | 24

2. Secondary Outcome: Percentage of Patients Who Were Normokalemic in the MP
Description: The percentage of patients who were normokalemic at each study visit in the MP is presented. Normokalemia was defined as a serum potassium (S-K) level of ≥ 3.5 and ≤ 5.0 mmol/L. The percentage of patients who were normokalemic at their last on-treatment visit is also presented. The last on-treatment value was defined as the last measurement taken within 1 day (2 days on QOD regimen) after the last ZS dose. End of Study was defined as the last ZS dose + 7 days.
Time Frame: MP Day 1 to End of Study visit (up to 12 months).
Population: The full analysis set for the MP (FAS-MP) included all patients who received at least 1 dose of ZS during the MP and who had any post-baseline MP S-K values.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Percentage of patients
  MP Day 1 | 82.0 [74.9 to 87.8]
  MP Day 2 | 78.7 [71.2 to 84.9]
  MP Day 5: number analyzed (Participants) | 149
  MP Day 5 | 79.9 [72.5 to 86.0]
  MP Day 12: number analyzed (Participants) | 149
  MP Day 12 | 67.8 [59.6 to 75.2]
  MP Day 19: number analyzed (Participants) | 148
  MP Day 19 | 65.5 [57.3 to 73.2]
  MP Day 26: number analyzed (Participants) | 148
  MP Day 26 | 72.3 [64.3 to 79.3]
  MP Day 54: number analyzed (Participants) | 144
  MP Day 54 | 76.4 [68.6 to 83.1]
  MP Day 82: number analyzed (Participants) | 140
  MP Day 82 | 72.1 [63.9 to 79.4]
  MP Day 110: number analyzed (Participants) | 137
  MP Day 110 | 75.9 [67.9 to 82.8]
  MP Day 138: number analyzed (Participants) | 134
  MP Day 138 | 85.1 [77.9 to 90.6]
  MP Day 166: number analyzed (Participants) | 132
  MP Day 166 | 78.0 [70.0 to 84.8]
  MP Day 194: number analyzed (Participants) | 130
  MP Day 194 | 75.4 [67.1 to 82.5]
  MP Day 222: number analyzed (Participants) | 129
  MP Day 222 | 70.5 [61.9 to 78.2]
  MP Day 250: number analyzed (Participants) | 129
  MP Day 250 | 79.8 [71.9 to 86.4]
  MP Day 278: number analyzed (Participants) | 127
  MP Day 278 | 75.6 [67.2 to 82.8]
  MP Day 306: number analyzed (Participants) | 124
  MP Day 306 | 74.2 [65.6 to 81.6]
  MP Day 334: number analyzed (Participants) | 124
  MP Day 334 | 83.1 [75.3 to 89.2]
  MP Day 362: number analyzed (Participants) | 122
  MP Day 362 | 79.5 [71.3 to 86.3]
  Last on-treatment Visit | 78.0 [70.5 to 84.3]
  End of Study Visit: number analyzed (Participants) | 146
  End of Study Visit | 38.4 [30.4 to 46.8]

3. Secondary Outcome: Percentage of Patients With Average S-K Levels of ≤5.1 mmol/L and ≤5.5 mmol/L in the MP
Description: The percentage of patients who had an average S-K level of ≤5.1 mmol/L and ≤5.5 mmol/L over the MP up to Day 362 is presented.
Time Frame: MP Day 2 to Day 362.
Population: The FAS-MP included all patients who received at least 1 dose of ZS during the MP and who had any post-baseline MP S-K values.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Percentage of patients
  ≤5.1 mmol/L | 93.3 [88.1 to 96.8]
  ≤5.5 mmol/L | 100.0 [97.6 to 100.0]

4. Secondary Outcome: Percentage of Patients Who Were Hypokalemic in the MP
Description: The percentage of patients who were hypokalemic at each study visit in the MP is presented. Hypokalemia was defined as a S-K level of < 3.5 mmol/L. The percentage of patients who were hypokalemic at their last on-treatment visit is also presented. The last on-treatment value was defined as the last measurement taken within 1 day (2 days on QOD regimen) after the last ZS dose. End of Study was defined as the last ZS dose + 7 days.
Time Frame: MP Day 1 to End of Study visit (up to 12 months).
Population: as for outcome 3
Measure: Number; unit: Percentage of patients
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Percentage of patients
  MP Day 1 | 0.0
  MP Day 2 | 0.0
  MP Day 5: number analyzed (Participants) | 149
  MP Day 5 | 0.0
  Day 12: number analyzed (Participants) | 149
  Day 12 | 0.0
  MP Day 19: number analyzed (Participants) | 148
  MP Day 19 | 0.0
  MP Day 26: number analyzed (Participants) | 148
  MP Day 26 | 0.7
  MP Day 54: number analyzed (Participants) | 144
  MP Day 54 | 2.8
  MP Day 82: number analyzed (Participants) | 140
  MP Day 82 | 3.6
  MP Day 110: number analyzed (Participants) | 137
  MP Day 110 | 0.7
  MP Day 138: number analyzed (Participants) | 134
  MP Day 138 | 2.2
  MP Day 166: number analyzed (Participants) | 132
  MP Day 166 | 1.5
  MP Day 194: number analyzed (Participants) | 130
  MP Day 194 | 0.8
  MP Day 222: number analyzed (Participants) | 129
  MP Day 222 | 1.6
  MP Day 250: number analyzed (Participants) | 129
  MP Day 250 | 2.3
  MP Day 278: number analyzed (Participants) | 127
  MP Day 278 | 1.6
  MP Day 306: number analyzed (Participants) | 124
  MP Day 306 | 1.6
  MP Day 334: number analyzed (Participants) | 124
  MP Day 334 | 1.6
  MP Day 362: number analyzed (Participants) | 122
  MP Day 362 | 1.6
  Last on-treatment Visit | 5.3
  End of Study Visit: number analyzed (Participants) | 146
  End of Study Visit | 0.7

5. Secondary Outcome: Percentage of Patients Who Were Hyperkalemic in the MP
Description: The percentage of patients who were hyperkalemic at each study visit in the MP is presented. Hyperkalemia was defined as a S-K level of >5.0 mmol/L. The percentage of patients who were hyperkalemic at their last on-treatment visit is also presented. The last on-treatment value was defined as the last measurement taken within 1 day (2 days on QOD regimen) after the last ZS dose. End of Study was defined as the last ZS dose + 7 days.
Time Frame: MP Day 1 to End of Study visit (up to 12 months).
Population: as for outcome 3
Measure: Number; unit: Percentage of patients
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Percentage of patients
  MP Day 1 | 18.0
  MP Day 2 | 21.3
  MP Day 5: number analyzed (Participants) | 149
  MP Day 5 | 20.1
  MP Day 12: number analyzed (Participants) | 149
  MP Day 12 | 32.2
  MP Day 19: number analyzed (Participants) | 148
  MP Day 19 | 34.5
  MP Day 26: number analyzed (Participants) | 148
  MP Day 26 | 27.0
  MP Day 54: number analyzed (Participants) | 144
  MP Day 54 | 20.8
  MP Day 82: number analyzed (Participants) | 140
  MP Day 82 | 24.3
  MP Day 110: number analyzed (Participants) | 137
  MP Day 110 | 23.4
  MP Day 138: number analyzed (Participants) | 134
  MP Day 138 | 12.7
  MP Day 166: number analyzed (Participants) | 132
  MP Day 166 | 20.5
  MP Day 194: number analyzed (Participants) | 130
  MP Day 194 | 23.8
  MP Day 222: number analyzed (Participants) | 129
  MP Day 222 | 27.9
  MP Day 250: number analyzed (Participants) | 129
  MP Day 250 | 17.8
  MP Day 278: number analyzed (Participants) | 127
  MP Day 278 | 22.8
  MP Day 306: number analyzed (Participants) | 124
  MP Day 306 | 24.2
  MP Day 334: number analyzed (Participants) | 124
  MP Day 334 | 15.3
  MP Day 362: number analyzed (Participants) | 122
  MP Day 362 | 18.9
  Last on-treatment Visit | 16.7
  End of Study Visit: number analyzed (Participants) | 146
  End of Study Visit | 61.0

6. Secondary Outcome: Mean Change From CP Baseline in the Mean S-K Level Over Specified Time Periods in the MP
Description: The mean changes from the CP baseline in S-K level over specified periods of time in the MP are presented. Baseline for the CP was defined as the mean of 2 different S-K values, recorded 60 minutes apart (to confirm qualification for study entry) on the CP Day 1.
Time Frame: CP Day 1 to MP Day 362.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
mmol/L
  MP Day 1 | -0.93 (0.44)
  Entire MP (Day 2 to Day 362) | -0.98 (0.42)
  MP Day 82 to Day 362: number analyzed (Participants) | 140
  MP Day 82 to Day 362 | -1.07 (0.52)
  MP Day 2 to Day 82 | -0.91 (0.41)
  MP Day 110 to Day 166: number analyzed (Participants) | 137
  MP Day 110 to Day 166 | -1.11 (0.61)
  MP Day 194 to Day 278: number analyzed (Participants) | 130
  MP Day 194 to Day 278 | -1.01 (0.51)
  MP Day 306 to Day 362: number analyzed (Participants) | 124
  MP Day 306 to Day 362 | -1.06 (0.55)

7. Secondary Outcome: Mean Change From MP Baseline in the Mean S-K Level Over Specified Time Periods in the MP
Description: The mean changes from the MP baseline in S-K level over specified periods of time in the MP are presented. Baseline for the MP was defined as the measurement taken in the morning of the day of entering the MP (MP Day 1).
Time Frame: MP Day 1 to Day 362.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
mmol/L
  Entire MP (Day 2 to Day 362) | -0.07 (0.33)
  MP Day 82 to Day 362: number analyzed (Participants) | 140
  MP Day 82 to Day 362 | -0.14 (0.42)
  MP Day 2 to Day 82 | -0.01 (0.36)
  MP Day 110 to Day 166: number analyzed (Participants) | 137
  MP Day 110 to Day 166 | -0.16 (0.50)
  MP Day 194 to Day 278: number analyzed (Participants) | 130
  MP Day 194 to Day 278 | -0.07 (0.42)
  MP Day 306 to Day 362: number analyzed (Participants) | 124
  MP Day 306 to Day 362 | -0.11 (0.47)

8. Secondary Outcome: Mean Number of Normokalemic Days During the MP
Description: The number of normokalemic days during the MP was calculated assuming the time interval between assessments was normokalemic if both the beginning and end assessments for that time interval displayed normal S-K values. If an intermediate scheduled assessment time point was missing, then the scheduled assessment was regarded as not normokalemic. The mean number of normokalemic days for a patient in the MP is presented.
Time Frame: MP Day 1 to Day 362.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Days | 207.7 (109.5)

9. Secondary Outcome: Mean Change in S-K Level From Last On-treatment MP Visit to the End of Study
Description: The mean change in the S-K level from the last on-treatment MP visit to the End of Study is presented. The last on-treatment value was defined as the last measurement taken within 1 day (2 days if on QOD regimen) after the last ZS dose. The End of Study was 7 days after the last ZS dose.
Time Frame: MP Day 1 to End of Study visit (up to 12 months).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
mmol/L | 0.66 (0.53)

10. Secondary Outcome: Change From CP Baseline in S-Aldosterone Levels Over the MP
Description: The mean change from CP baseline to MP Day 166 and MP Day 362 in S-aldosterone levels is presented. In addition, the mean change from CP baseline to the last on-treatment value is presented. The CP baseline was defined as the last S-aldosterone assessment immediately prior to the start of the first dose of ZS during the CP. The last on-treatment value was defined as the last measurement taken within 1 day (2 days if on QOD regimen) after the last ZS dose.
Time Frame: CP Day 1, MP Day 166 and MP Day 362.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Picomole per liter (pmol/L)
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Picomole per liter (pmol/L)
  MP Day 166: number analyzed (Participants) | 131
  MP Day 166 | -56.355 (124.050)
  MP Day 362: number analyzed (Participants) | 121
  MP Day 362 | -48.561 (129.261)
  Last on-treatment Visit: number analyzed (Participants) | 131
  Last on-treatment Visit | -48.808 (125.081)

11. Secondary Outcome: Percentage of Patients With Normal S-Aldosterone Levels Over the MP
Description: The percentage of patients with normal S-aldosterone levels up to Day 362 of the MP is presented. The normal range for S-aldosterone was 0 - 776.72 pmol/L. In addition, the percentage of patients with normal S-aldosterone levels at the last on-treatment visit is presented. The CP baseline was defined as the last S-aldosterone assessment immediately prior to the start of the first dose of ZS during the CP. The last on-treatment value was defined as the last measurement taken within 1 day (2 days if on QOD regimen) after the last ZS dose.
Time Frame: CP Day 1, MP Day 166 and MP Day 362.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Percentage of patients
  CP Baseline: number analyzed (Participants) | 148
  CP Baseline | 99.3 [96.3 to 100.0]
  MP Day 166: number analyzed (Participants) | 132
  MP Day 166 | 100.0 [97.2 to 100.0]
  MP Day 362: number analyzed (Participants) | 122
  MP Day 362 | 100.0 [97.0 to 100.0]
  Last on-treatment Visit: number analyzed (Participants) | 132
  Last on-treatment Visit | 100.0 [97.2 to 100.0]

12. Secondary Outcome: Change From CP Baseline in S-Bicarbonate Levels Over the MP
Description: The mean change from CP baseline to timepoints in the MP in S-bicarbonate levels is presented. In addition, the mean change from CP baseline to the last on-treatment value is presented. The CP baseline was defined as the last S-bicarbonate assessment immediately prior to the start of the first dose of ZS during the CP. The last on-treatment value was defined as the last measurement taken within 1 day (2 days if on QOD regimen) after the last ZS dose. The End of Study was 7 days after the last ZS dose.
Time Frame: CP Day 1, and MP Day 1 to End of Study visit (up to 12 months).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
mmol/L
  MP Day 1: number analyzed (Participants) | 148
  MP Day 1 | 1.20 (1.64)
  MP Day 5: number analyzed (Participants) | 148
  MP Day 5 | 1.20 (1.71)
  MP Day 12: number analyzed (Participants) | 147
  MP Day 12 | 1.46 (1.91)
  MP Day 19: number analyzed (Participants) | 147
  MP Day 19 | 1.29 (2.27)
  MP Day 26: number analyzed (Participants) | 148
  MP Day 26 | 1.64 (2.22)
  MP Day 82: number analyzed (Participants) | 139
  MP Day 82 | 1.45 (2.90)
  MP Day 166: number analyzed (Participants) | 132
  MP Day 166 | 1.55 (2.53)
  MP Day 250: number analyzed (Participants) | 129
  MP Day 250 | 1.84 (2.64)
  MP Day 334: number analyzed (Participants) | 124
  MP Day 334 | 1.73 (2.75)
  MP Day 362: number analyzed (Participants) | 122
  MP Day 362 | 1.50 (2.85)
  Last on-treatment Visit | 1.70 (2.87)
  End of Study Visit: number analyzed (Participants) | 146
  End of Study Visit | 0.55 (2.49)

13. Secondary Outcome: Percentage of Patients With Normal S-Bicarbonate Levels Over the MP
Description: The percentage of patients with normal S-bicarbonate levels up to the End of Study visit in the MP is presented. The normal range for S-bicarbonate was 17 - 32 mmol/L. In addition, the percentage of patients with normal S-bicarbonate levels at the last on-treatment visit is presented. The CP baseline was defined as the last S-bicarbonate assessment immediately prior to the start of the first dose of ZS during the CP. The last on-treatment value was defined as the last measurement taken within 1 day (2 days if on QOD regimen) after the last ZS dose. The End of Study was 7 days after the last ZS dose.
Time Frame: CP Day 1 and MP Day 1 to End of Study visit (up to 12 months).
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Percentage of patients
  CP Baseline | 90.0 [84.0 to 94.3]
  MP Day 1: number analyzed (Participants) | 148
  MP Day 1 | 98.0 [94.2 to 99.6]
  MP Day 5: number analyzed (Participants) | 148
  MP Day 5 | 98.6 [95.2 to 99.8]
  MP Day 12: number analyzed (Participants) | 147
  MP Day 12 | 98.0 [94.2 to 99.6]
  MP Day 19: number analyzed (Participants) | 147
  MP Day 19 | 97.3 [93.2 to 99.3]
  MP Day 26: number analyzed (Participants) | 148
  MP Day 26 | 98.6 [95.2 to 99.8]
  MP Day 82: number analyzed (Participants) | 139
  MP Day 82 | 97.8 [93.8 to 99.6]
  MP Day 166: number analyzed (Participants) | 132
  MP Day 166 | 99.2 [95.9 to 100.0]
  MP Day 250: number analyzed (Participants) | 129
  MP Day 250 | 99.2 [95.8 to 100.0]
  MP Day 334: number analyzed (Participants) | 124
  MP Day 334 | 97.6 [93.1 to 99.5]
  MP Day 362: number analyzed (Participants) | 122
  MP Day 362 | 95.9 [90.7 to 98.7]
  Last on-treatment Visit | 96.7 [92.4 to 98.9]
  End of Study Visit: number analyzed (Participants) | 146
  End of Study Visit | 93.8 [88.6 to 97.1]

14. Secondary Outcome: Baseline and Post-baseline 36-Item Short Form Health Survey Version 2 (SF-36 v2) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: Patients completed the SF-36 v2 questionnaire on Day 1 of the CP and on Day 362 of the MP. The responses to the items assessing the physical and mental health of the patients determined the PCS and MCS based on a standard algorithm. The PCS and MCS scores ranged from 0 (worst possible health state) to 100 (best possible health state). The mean PCS and MCS are presented for the baseline and post-baseline assessments.
Time Frame: CP Day 1 (baseline) and MP Day 362 (post-baseline).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Scale score
  Baseline: PCS | 49.106 (6.292)
  Post-baseline: PCS: number analyzed (Participants) | 127
  Post-baseline: PCS | 49.348 (6.659)
  Baseline: MCS | 51.126 (8.375)
  Post-baseline: MCS: number analyzed (Participants) | 127
  Post-baseline: MCS | 50.350 (8.384)

15. Secondary Outcome: Mean Change From CP Baseline in the Mean S-K Levels in the CP
Description: The mean change from the CP baseline at 24, 48 and 72 hours in the CP is presented. The mean change from baseline to the last on-treatment CP value is also presented. The last on-treatment value was defined as the last measurement taken with 1 day (2 days if on the QOD regimen) after the last ZS dose. Baseline for the CP was defined as the mean of 2 different S-K values, recorded 60 minutes apart (to confirm qualification for study entry) on the CP Day 1.
Time Frame: CP Day 1 to Day 3.
Population: The CP full analysis set (FAS-CP) included all patients who received at least 1 dose of ZS during the CP and who had any post-baseline CP S-K values.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
mmol/L
  24 hours | -0.78 (0.39)
  48 hours: number analyzed (Participants) | 32
  48 hours | -1.30 (0.39)
  72 hours: number analyzed (Participants) | 1
  72 hours | NA (NA) — Data for a single patient not reported for data privacy reasons.
  Last on-treatment Visit | -0.93 (0.44)

16. Secondary Outcome: Percentage of Patients Who Were Normokalemic in the CP
Description: The percentage of patients who were normokalemic at 24, 48 and 72 hours in the CP is presented. Normokalemia was defined as a S-K level of ≥ 3.5 and ≤ 5.0 mmol/L.
Time Frame: CP Day 1 to Day 3.
Population: The FAS-CP included all patients who received at least 1 dose of ZS during the CP and who had any post-baseline CP S-K values.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Percentage of patients
  24 hours | 65.3 [57.1 to 72.9]
  48 hours | 81.3 [74.2 to 87.2]
  72 hours: number analyzed (Participants) | 149
  72 hours | 82.0 [74.9 to 87.8]

17. Secondary Outcome: Number of Patients Who Experienced AEs in the CP
Description: The number of patients who experienced any AE, including SAEs, those which had an outcome of death, were severe, led to discontinuation of ZS or were causally related to ZS are presented for the CP. AEs of special interest are also presented, including oedema-related AEs, cardiac failure and hypertension.
Time Frame: Day 1 of CP to last CP dose + 1 day or first MP dose -1 day, earlier.
Population: The SAF-CP included all patients treated with at least 1 dose of CP ZS and who had any CP safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate
Number analyzed (Participants) | 150
Participants
  Any AE | 5
  Any AE with outcome death | 0
  Any SAE | 1
  Any severe AE | 0
  Any AE leading to ZS discontinuation | 0
  Any causally related AE | 0
  Oedema-related AE | 0
  Cardiac failure | 0
  Hypertension | 0

ADVERSE EVENTS:
Time Frame: For the CP, from Day 1 to last CP dose + 1 day or first MP dose -1 day. For the MP, from the first MP dose up to 1 day (2 days for QOD regimen) after last MP dose. Overall, approximately 12 months.
Description: AE data is presented for the SAF-MP which included all patients treated with at least 1 dose of MP ZS and had any MP safety data, and for the SAF-CP which included all patients treated with at least 1 dose of CP ZS and had any CP safety data.
Groups:
- Correction Phase: CP (up to 3 days):
  Patients received 10 g ZS TID for a maximum of 72 hours.
- Maintenance Phase: MP (up to 12 months):
  Patients received a starting dose of 5 g ZS QD which could be increased to 10 g or 15 g QD or decreased to 5 g QOD or 2.5 g QD.
Arm/Group | Correction Phase | Maintenance Phase
All-Cause Mortality (participants affected / at risk) | 0/150 | 2/150
Serious Adverse Events (participants affected / at risk) | 1/150 | 27/150
Other Adverse Events (participants affected / at risk) | 1/150 | 79/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Correction Phase (N=150) | Maintenance Phase (N=150)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Pyelonephritis (Infections and infestations) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Undifferentiated sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Diabetic retinopathy (Eye disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 1
Strabismus (Eye disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 4
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Correction Phase (N=150) | Maintenance Phase (N=150)
Oedema peripheral (General disorders) | 0 | 23
Nasopharyngitis (Infections and infestations) | 1 | 36
Hypertension (Vascular disorders) | 0 | 23
Constipation (Gastrointestinal disorders) | 0 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT03172702/SAP_000.pdf
  • Study Protocol (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT03172702/Prot_001.pdf